CLINICAL TRIAL: NCT04596540
Title: A Randomized Double-Blind, Placebo-Controlled Study of SEL-212 in Patients With Gout Refractory to Conventional Therapy
Brief Title: A Study of SEL-212 in Patients With Gout Refractory to Conventional Therapy II
Acronym: DISSOLVE II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEL-212/302; 2020-003070-45 (EudraCT Number)
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Chronic Gout

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SEL-212 low-dose (Experimental): IV infusion of SEL-212 low-dose every 28 days for a total of up to 6 infusions
  Interventions: Drug: SEL-212 low-dose
- SEL-212 high-dose (Experimental): IV infusion of SEL-212 high-dose every 28 days for a total of up to 6 infusions
  Interventions: Drug: SEL-212 high-dose
- Placebo (Placebo Comparator): IV infusion of Normal Saline every 28 days for a total of up to 6 infusions
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SEL-212 low-dose — SEL-212 low-dose Drug: SEL-037 (0.2 mg/kg) SEL-037, PEGylated uric acid specific enzyme (uricase) Other Names: Pegadricase, pegsiticase
  Drug: SEL-110.36 (0.1 mg/kg) Other Names: SEL-110, ImmTOR
  Arms: SEL-212 low-dose
Drug: SEL-212 high-dose — SEL-212 high-dose Drug: SEL-037 (0.2 mg/kg) SEL-037, PEGylated uric acid specific enzyme (uricase) Other Names: Pegadricase, pegsiticase
  Drug: SEL-110.36 (0.15 mg/kg) Other Names: SEL-110, ImmTOR
  Arms: SEL-212 high-dose
Other: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
This is one of two replicate randomized, double-blind, placebo-controlled, parallel arm trials to determine the safety and efficacy of two different dose levels of SEL-212 compared to placebo. 112 and 153 patients, stratified as to the presence or absence of tophi, were randomized in a 1:1:1 allocation ratio prior to Baseline to receive treatment with one of two dose levels of SEL-212 or placebo every 28 days for approximately 6 months in each trial respectively (SEL-212/301 and SEL-212/302). Analysis of primary and key efficacy were performed at Day 28 of Treatment Period 6. Safety was monitored throughout the study.

DETAILED DESCRIPTION:
This is one of two replicate randomized, double-blind, placebo-controlled, parallel arm trials to determine the safety and efficacy of two different dose levels of SEL-212 compared to placebo. 112 and 153 patients, stratified as to the presence or absence of tophi, were randomized in a 1:1:1 allocation ratio prior to Baseline to receive treatment with one of two dose levels of SEL-212 or placebo every 28 days for approximately 6 months in each trial respectively (SEL-212/301 and SEL-212/302). The SEL-212 doses differed as to the SEL-110.36 component. Participants received SEL-037 administered at a dose of 0.2 mg/kg via intravenous (IV) infusion immediately after receiving SEL-110.36 at a dose of either 0.1 mg/kg (SEL-212 low-dose) or 0.15 mg/kg (SEL-212 high-dose) via IV infusion. The placebo consisted of normal saline.

Efficacy assessments were conducted at intervals that are appropriate to determine treatment effect with samples for the primary endpoint drawn during Treatment Period 6. Safety was monitored throughout the study with an independent data safety monitoring board (DSMB).

ELIGIBILITY:
Inclusion Criteria:

1. Has negative results of an FDA Emergency Use Authorized COVID-19 molecular assay for detection of SARS-CoV-2 RNA from a nasal or oropharyngeal specimen;
2. History of symptomatic gout defined as:

   1. ≥ 3 gout flares within 18 months of Screening or
   2. Presence of ≥ 1 gout tophus or
   3. Current diagnosis of gouty arthritis
3. At the Screening Visit: male age 21 - 80 years, inclusive, or female of non-childbearing potential age 21-80 years, inclusive, where nonchildbearing potential is defined as:

   1. > 6 weeks after hysterectomy with or without surgical bilateral salpingo-oophorectomy or
   2. Post-menopausal (> 24 months of natural amenorrhea or in the absence of >24 months of amenorrhea, one documented confirmatory FSH measurement)
4. Has chronic refractory gout defined as having failed to normalize sUA and whose signs and symptoms are inadequately controlled with any of the xanthine oxidase inhibitors, or for whom these drugs are contraindicated for the patient;
5. Has at the Screening Visit SUA ≥ 7 mg/dL
6. Negative serology for HIV-1/-2 and negative antigen to hepatitis B and negative antibodies to hepatitis C;

Exclusion Criteria:

1. Has a history of anaphylaxis, severe allergic reactions, or severe atopy;
2. Has a history of any allergy to pegylated products, including, but not limited to pegloticase (Krystexxa®), peginterferon alfa-2a (Pegasys®), peginterferon alfa-2b (PegIntron®), pegfilgrastim (Neulasta®), pegaptanib (Macugen®), pegaspargase (Oncaspar®), pegademase (Adagen®), peg-epoetin beta (Mircera®), pegvisomant (Somavert®) certolizumab pegol (Cimzia®), naloxegol (Movantik®), peginesatide (Omontys®), and doxorubicin liposome (Doxil®);
3. Is taking and cannot discontinue known major CYP3A4/P-gp inhibitors or major CYP3A4/P-gp inducers at least 14 days before dosing. Patients must remain off these medications for the duration of the study, including natural products such as St. John's Wort or grapefruit juice.
4. Is taking drugs known to interact with rapamycin (sirolimus - Rapamune®) such as cyclosporine, diltiazem, erythromycin, ketoconazole, posaconazole, voriconazole, itraconazole, rifampin, verapamil unless they are stopped 14 days prior to dosing and will not be used/prescribed during the trial.
5. Had major surgery within 3 months of initial screening.
6. Had a gout flare during Screening that was resolved for less than 1 week prior to first treatment with study drug (exclusive of chronic synovitis/arthritis) unless the patient has a history of inter-flare intervals of < 1 week.
7. Has uncontrolled diabetes at Screening with HbA1c ≥ 8.5%;
8. Has fasting Screening glucose > 240 mg/dL;
9. Has fasting Screening triglyceride > 500 mg/dL;
10. Has fasting Screening low-density lipoprotein (LDL) > 200 mg/dL;
11. Has glucose-6-phosphate dehydrogenase (G6PD) deficiency;
12. Has uncontrolled hypertension defined as blood pressure > 170/100 mmHg at Screening and 1 week prior to dosing
13. Individual laboratory values which are exclusionary

    * White blood cell count (WBC) < 3.0 x109/L
    * Serum aspartate aminotransferase (AST) or alanine amino transferase (ALT) > 3x upper limit of normal (ULN) in the absence of known active liver disease
    * Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2
    * Urine albumin creatinine ratio (UACR) > 30 mg/g
    * Hemoglobin (Hgb) < 9 g/dL
    * Serum phosphate < 2.0 mg/dL
14. Is receiving ongoing treatment for arrhythmia, including placement of an implantable defibrillator, unless considered stable and on active treatment;
15. Has evidence of unstable cardiovascular disease or unstable cerebrovascular vascular disease. This includes patients who have had a cardiac/vascular event(s) in the last 3 months including heart attack, stroke or vascular bypass surgery or patients who are deemed, by their physician or PI, to have active cardiovascular, cerebrovascular or peripheral vascular symptoms/disease inadequately controlled by medication;
16. Has congestive heart failure, New York Heart Association Class III or IV;
17. Unless clinically stable and/or appropriately treated, electrocardiogram (ECG) with evidence of clinically significant arrhythmia or other abnormalities that, in the opinion of the investigator, are consistent with significant underlying cardiac disease;
18. History of significant hematological disorders within 5 years or autoimmune disorders, and/or patient is currently immunosuppressed or immunocompromised;
19. Prior exposure to any experimental or marketed uricase (e.g., rasburicase (Elitek, Fasturtec), pegloticase (Krystexxa®®), pegadricase (SEL 037))
20. Patient has received a live vaccine in the previous 6 months.
21. Patient is planning to receive any live vaccine during the study.
22. History of malignancy within the last 5 years other than basal skin cancer;
23. Patients with a documented history of moderate or severe alcohol or substance use disorder within the 12 months prior to randomization.
24. History of or evidence of clinically severe interstitial lung disease
25. Immunocompromised state, regardless of etiology

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female of non-childbearing potential defined as either >6 weeks after hysterectomy with or without surgical bilateral salpingo-oophorectomy OR post-menopausal (> 24 months of natural amenorrhea or in the absence of > 24 months of amenorrhea, one documented confirmatory FSH measurement)
Enrollment: 153 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Swedish Orphan Biovitrum AB (publ)
Locations (53):
- United States (30):
  - Clinical Research Of West Florida Incorporated, Clearwater, Florida
  - Omegas Research Consultants LLC, DeBary, Florida
  - Sweet Hope Research Specialty, Inc, Hialeah, Florida
  - Homestead Associates in Research,Inc, Miami, Florida
  - D&H National Research Centers, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Napa Research, Pompano Beach, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Horizon Clinical Research, Fayetteville, Georgia
  - Arthritis Center of North Georgia, LLC, Gainesville, Georgia
  - Injury Care Medical Center, Boise, Idaho
  - Great Lakes Clinical Trials at Ravenswood Rheumatology, Chicago, Illinois
  - Great Lakes Clinical Trials LLC, Chicago, Illinois
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - University Of Michigan, Ann Arbor, Michigan
  - Elite Clinical Research, LLC, Jackson, Mississippi
  - Rutgers- New Jersey Medical School, Newark, New Jersey
  - Medication Management of Greensboro, Greensboro, North Carolina
  - Triad Clinical Trials, Greensboro, North Carolina
  - Carolina Research Center, Inc, Shelby, North Carolina
  - META Medical Research Institute LLC, Dayton, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - New Phase Research and Development, Knoxville, Tennessee
  - Amarillo Center for Clinical Research, Ltd., Amarillo, Texas
  - Heritage Rheumatology and Arthritis Care, Colleyville, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Southwest Rheumatology Research LLC, Mesquite, Texas
  - AIM Trials - Internal Medicine, Plano, Texas
  - Arthritis Northwest, PLLC - Research, Spokane, Washington
- Georgia (6):
  - Aleksandre Aladashvili Clinic LLC, Tbilisi
  - LTD Israeli-Georgian Medical Research Clinic "Helsicore", Tbilisi
  - JSC "Evex Hospitals", Tbilisi
  - LTD MediClub Georgia, Tbilisi
  - LTD Georgian-Dutch Hospital, Tbilisi
  - LTD "The First Medical Center", Tbilisi
- Russia (6):
  - Republican Hospital n.a. V.A. Baranov, Petrozavodsk, Kareliya, Respublika
  - Research Institute of Rheumatology n.a. Nasonova, Moscow, Moscow
  - GBOU VPO Orenburg State Medical University, Orenburg, Orenburg Oblast
  - Ryazan State Medical University n. a. I.P. Pavlov, Ryazan, Ryazan Oblast
  - Clinical Rheumatological Hospital #25, Saint Petersburg, Sankt-Peterburg
  - Medical-sanitary unit #157 - Rheumatology, Saint Petersburg, Sankt-Peterburg
- Serbia (5):
  - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja, Nišavski Okrug
  - Institute for Rheumatology - Rheumatology, Belgrade
  - Institute for Rheumatology, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Hospital Center Bezanisjka Kosa, Belgrade
- Ukraine (6):
  - Tovarystvo z obmezhenoi vidpov, Kyiv, Kyïv
  - Naukovo-Doslidnyi Inst. Reabil, Vinnytsia, Vinnytsia Oblast
  - Medychnyi tsentr Tovarystva z, Zaporizhzhia, Zaporizhzhia Oblast
  - Cherkaska Oblasna likarnia, Cherkasy
  - Kyivska klinichna likarnia na, Kyiv
  - Vinnytska Oblasna klinichna likarnia imeni M.I, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SEL-212A (Low-dose): SEL-212 is comprised of 2 components: SEL-037 and SEL-110. Participants received SEL-037 administered at a dose of 0.2 milligrams per kilogram (mg/kg) via intravenous (IV) infusion immediately after receiving SEL-110 at a dose of 0.1 mg/kg (SEL-212A) every 28 days for approximately six months.
- SEL-212B (High-dose): SEL-212 is comprised of 2 components: SEL-037 and SEL-110. Participants received SEL-037 administered at a dose of 0.2 mg/kg via IV infusion immediately after receiving SEL-110 at a dose of 0.15 mg/kg (SEL-212B) every 28 days for approximately six months.
- Placebo: Participants received placebo (normal saline) via IV infusion every 28 days for approximately six months.
Period: Overall Study
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Started | 51 | 49 | 53
Received at Least 1 Dose of Study Treatment | 51 | 49 | 53
Completed | 33 | 33 | 44
Not Completed | 18 | 16 | 9
Not completed — Withdrawal by Subject | 9 | 8 | 5
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Sponsor Decision | 2 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Coronavirus Disease 2019 (COVID-19) | 1 | 0 | 0
Not completed — Other Than Specified | 5 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Safety Set, which included all participants who were administered any amount of study medication. Participants were analyzed according to treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo | Total
Number analyzed (Participants) | 51 | 49 | 53 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.60) | 56.4 (9.70) | 56.5 (10.05) | 55.4 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 49 | 47 | 52 | 148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 1 | 4
  Not Hispanic or Latino | 48 | 49 | 52 | 149
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 8 | 15
  White | 45 | 47 | 44 | 136
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Achieved and Maintained Reduction in Serum Uric Acid (sUA) < 6 Milligrams Per Deciliter (mg/dL) for At Least 80% of The Time During Treatment Period 6 (Month 6)
Time Frame: Month 6
Population: The Intent-to-Treat (ITT) Set, which included all randomized and dosed participants, including participants with missing data that were multiple imputed. Participants were analyzed according to randomized treatment.
Measure: Number; unit: proportion of participants
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 51 | 49 | 53
proportion of participants | 0.40 | 0.46 | 0.11
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p = 0.0008, Mantel Haenszel; Risk Difference (RD) = 0.29, 97.5% CI 2-sided [0.10 to 0.48]
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p = 0.0002, Mantel Haenszel; Risk Difference (RD) = 0.35, 97.5% CI 2-sided [0.14 to 0.56]

2. Secondary Outcome: Change From Baseline in Mean sUA
Time Frame: Baseline up to 6 months
Population: The ITT Set, which included all randomized and dosed participants including participants with missing data that were multiple imputed. Participants were analyzed according to randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 51 | 49 | 53
milligrams per deciliter (mg/dL) | -4.0 (0.6) | -5.1 (0.6) | -0.6 (0.5)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Least Squares (LS) Mean Difference = -3.3, 97.5% CI 2-sided [-5.07 to -1.55], Standard Error of Mean 0.8
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -4.5, 97.5% CI 2-sided [-6.24 to -2.66], Standard Error of Mean 0.8

3. Secondary Outcome: Percentage Change From Baseline in Mean sUA
Time Frame: Baseline up to 6 months
Population: The ITT Set, which included all randomized and dosed participants, including participants with missing data that were multiple imputed. Participants were analyzed according to randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 51 | 49 | 53
percentage change | -46.3 (6.9) | -59.8 (7.3) | -6.2 (6.3)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p < .001, ANCOVA; LS Mean Difference = -40.1, 97.5% CI 2-sided [-60.96 to -19.27], Standard Error of Mean 9.3
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p < .001, ANCOVA; LS Mean Difference = -53.6, 97.5% CI 2-sided [-74.49 to -32.66], Standard Error of Mean 9.3

4. Secondary Outcome: Change From Baseline in the Physical Component Summary Score of the Short Form Health Survey (SF-36)
Description: The SF-36 is a 36-item scale constructed to survey health status and quality of life (QoL). The SF-36 assesses 8 health concepts, which are the weighted sums of the questions in their section: limitations in physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems; bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions. Each scale was directly transformed into a 0-100 scale, and the total average scores were calculated across the 8 health concepts. The 8 domains contribute to physical component summary and mental component summary scores. Total scores for the physical component summary score ranged from 0-100, with a higher score indicating better health outcomes.
Time Frame: Baseline up to 6 months
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 51 | 49 | 53
scores on a scale | 10.4 (1.4) | 8.4 (1.3) | 3.8 (1.2)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean Difference = 6.6, 97.5% CI 2-sided [2.52 to 10.66], Standard Error of Mean 1.8
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p = 0.011, Mixed Models Analysis; LS Mean Difference = 4.6, 97.5% CI 2-sided [0.54 to 8.59], Standard Error of Mean 1.8

5. Secondary Outcome: Proportion of Participants With at Least Partial Response (PR) (as Best Response) in Overall Tophus Response Evaluation in Participants With Tophi at Baseline
Description: Baseline photographs of the hands and feet of each participant were obtained using a standardized method in all participants, together with photographs of up to two other representative sites of tophaceous disease. The baseline photographs were assessed by three independent reviewers to prospectively identify sites of tophaceous disease present at the start of treatment. Up to five tophi in the photographs were chosen by the reviewers for measurement over the course of therapy. The reviewers assessed the photographs for size of each target tophus using image analysis software. At least PR was defined as at least a 50% decrease in the area of at least one tophus, and includes participants with complete response (CR). Data are presented for the proportion of participants with at least PR (as best response) in overall tophus response evaluation.
Time Frame: Baseline Up to 6 months
Population: The ITT Set, which included all randomized and dosed participants, including participants with missing data that were multiple imputed. Participants were analyzed according to randomized treatment. Here, overall number of participants analyzed = participants with tophi at baseline with evaluable data for the outcome measure.
Measure: Number (97.5% Confidence Interval); unit: proportion of participants
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 34 | 33 | 36
proportion of participants | 0.83 [0.81 to 0.85] | 0.93 [0.91 to 0.94] | 0.54 [0.52 to 0.56]
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p = 0.0470, Chi-squared; Difference = 0.30, 97.5% CI 2-sided [-0.02 to 0.62]
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p = 0.0022, Chi-squared; Difference = 0.39, 97.5% CI 2-sided [0.12 to 0.66]

6. Secondary Outcome: Proportion of Participants Who Achieved and Maintained Reduction of sUA < 6 mg/dL for at Least 80% of the Time During Month 6 in the Subset of Participants With Tophi at Baseline
Description: The number of responders in the subgroup of ITT participants with tophi at baseline divided by the number of ITT participants with tophi at baseline.
Time Frame: Baseline up to 6 months
Population: as for outcome 5
Measure: Number (97.5% Confidence Interval); unit: proportion of participants
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 34 | 33 | 36
proportion of participants | 0.38 [0.38 to 0.39] | 0.45 [0.44 to 0.47] | 0.11 [0.10 to 0.11]
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p = 0.0096, Chi-squared; Difference = 0.28, 97.5% CI 2-sided [0.05 to 0.51]
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p = 0.0028, Chi-squared; Difference = 0.35, 97.5% CI 2-sided [0.10 to 0.60]

7. Secondary Outcome: Change From Baseline to Month 6 in Number of Tender Joints
Description: Tender and/or swollen joints were counted. The following joints were assessed: metacarpophalangeal, proximal interphalangeal, and distal interphalangeal joints of the hands; the metatarsophalangeal and interphalangeal joints of the feet; shoulder, elbow, wrist, knee, ankle, tarsus, sternoclavicular, and acromioclavicular joints. Data are presented for the mean change from baseline in number of tender joints.
Time Frame: Baseline up to 6 months
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: tender joints
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 51 | 49 | 53
tender joints | -9.2 (0.9) | -8.1 (0.9) | -4.4 (0.8)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean Difference = -4.8, 97.5% CI 2-sided [-7.55 to -1.98], Standard Error of Mean 1.2
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis; LS Mean Difference = -3.7, 97.5% CI 2-sided [-6.42 to -0.91], Standard Error of Mean 1.2

8. Secondary Outcome: Change From Baseline to Month 6 in the Total Score of the Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ-DI assesses fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both the upper and lower extremities. It includes 20 items in 8 categories: "activity", "arising", "dressing and grooming", "eating", "grip", "hygiene", "reach", and "walking". Scoring within each section was on a 4-point Likert scale from 0 (without any difficulty) to 3 (unable to do), with higher scores showing more disability. The average of the 8 category scores was reported as the HAQ-DI total score on a scale of 0 to 3, with higher scores showing more disability. Data are reported for change from baseline to Month 6 in the total HAQ-DI score. A decrease in HAQ-DI score from baseline indicated an improvement in the participant's condition.
Time Frame: Baseline up to 6 months
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 51 | 49 | 53
scores on a scale | -0.6 (0.1) | -0.4 (0.1) | -0.3 (0.1)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p = 0.018, Mixed Models Analysis; LS Mean Difference = -0.2, 97.5% CI 2-sided [-0.46 to -0.01], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p = 0.785, Mixed Models Analysis; LS Mean Difference = 0.0, 97.5% CI 2-sided [-0.25 to 0.20], Standard Error of Mean 0.1

9. Secondary Outcome: Incidence of Gout Flare During Treatment Periods 1-6 (Months 1-6)
Description: Gout flare was assessed as part of adverse event (AE) collection. Gout flares were assessed during the Treatment Phase using a validated definition of flares in participants with established gout. A gout flare (per Gaffo et al. 2018) was defined as the fulfilment of at least 3 of the following 4 criteria: 1. Participant-defined gout flare, 2. Pain at rest score of >3 on a 0-10-point numerical rating scale, 3. Presence of at least 1 swollen joint, 4. Presence of at least 1 warm joint. Data are presented for the mean incidence per month of gout flares during Treatment Periods 1-6 (Months 1-6). A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Months 1-6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: gout flares/month
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 51 | 49 | 53
gout flares/month | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p = 0.500, ANOVA; LS Mean Difference = 0.0, 97.5% CI 2-sided [-0.15 to 0.08]
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p = 0.421, ANOVA; LS Mean Difference = 0.0, 97.5% CI 2-sided [-0.15 to 0.07]

10. Secondary Outcome: Incidence of Gout Flare During Treatment Periods 1-3 (Months 1-3)
Description: Gout flare was assessed as part of adverse event (AE) collection. Gout flares were assessed during the Treatment Phase using a validated definition of flares in participants with established gout. A gout flare (per Gaffo et al. 2018) was defined as the fulfilment of at least 3 of the following 4 criteria: 1. Participant-defined gout flare, 2. Pain at rest score of >3 on a 0-10-point numerical rating scale, 3. Presence of at least 1 swollen joint, 4. Presence of at least 1 warm joint. Data are presented for the mean incidence per month of gout flares during Treatment Periods 1-3 (Months 1-3). A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Months 1-3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: gout flares/month
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 51 | 49 | 53
gout flares/month | 0.1 (0.1) | 0.2 (0.1) | 0.2 (0.1)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Treatment Periods 1-3 (Months 1-3); Test type: Superiority; p = 0.634, ANOVA; LS Mean Difference = 0.0, 97.5% CI 2-sided [-0.22 to 0.14], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Treatment Periods 1-3 (Month 1-3); Test type: Superiority; p = 0.907, ANOVA; LS Mean Difference = 0.0, 97.5% CI 2-sided [-0.17 to 0.19], Standard Error of Mean 0.1

ADVERSE EVENTS:
Time Frame: Up to approximately 6 months
Description: Safety Set, which included all participants who were administered any amount of study drug. Participants were analyzed according to treatment received.
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49 | 0/53
Serious Adverse Events (participants affected / at risk) | 5/51 | 4/49 | 2/53
Other Adverse Events (participants affected / at risk) | 28/51 | 26/49 | 27/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SEL-212A (Low-dose) (N=51) | SEL-212B (High-dose) (N=49) | Placebo (N=53)
COVID-19 (Infections and infestations) | 0 | 0 | 1
Infected gouty tophus (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SEL-212A (Low-dose) (N=51) | SEL-212B (High-dose) (N=49) | Placebo (N=53)
Gout (Metabolism and nutrition disorders) | 18 | 18 | 18
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 3
Dyslipidaemia (Metabolism and nutrition disorders) | 3 | 3 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 4
COVID-19 (Infections and infestations) | 2 | 3 | 4
Nasopharyngitis (Infections and infestations) | 0 | 2 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 3 | 0
Hypertension (Vascular disorders) | 0 | 3 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0
Microalbuminuria (Renal and urinary disorders) | 1 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT04596540/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT04596540/SAP_001.pdf